CLINICAL TRIAL: NCT07147166
Title: Evaluating the Efficacy of Force Modulating Tissue Bridge Device in Preventing Hypertrophic Scars Following Gender-Affirming Mastectomy: A Randomized Self-Controlled Trial
Brief Title: Evaluating the Efficacy of Force Modulating Tissue Bridge Device in Preventing Hypertrophic Scars Following Gender-Affirming Mastectomy
Acronym: FMTB Brij
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Esther Kim, MD, Esther A. Kim, MD, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-43094
Record Dates: First submitted 2025-07-29; First posted 2025-08-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-08

CONDITIONS: Gender Dysphoria; Mastectomy; Hypertrophic Scar
Keywords: Gender-affirming; Gender-affirming care; Gender-affirming mastectomy; Hypertrophic scarring
MeSH Terms: conditions — Gender Dysphoria; Cicatrix, Hypertrophic

STUDY DESIGN:
Masking Description: While study participants cannot be blinded to the intervention, the operating surgeon will remain blinded to the patient's assignment until final skin closure at the end of the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Self-control Brijjit Application and Control (Experimental): The side of the chest that the Brijjit is applied to will be randomly allocated using a web-based, open-source randomizer. Initial application will be done intraoperatively, following final skin closure. Brijjit will be applied across the entire incision length. Following application, Brijjit has been shown to last for 2-4 weeks. Patients will remain in a chest vest binder with dressings until the initial follow-up visit at 2 weeks. At this follow up visit, any Brijjit that has fallen off will be replaced. Patients will be taught how to reapply Brijjit if it falls off, and they will be instructed to continue Brijjit therapy until 6 weeks post-op. Any remaining Brijjit devices will be removed at the 6 week post-op visit. At this time, patients will be able to initiate recommended scar care to both chest sides.
  The control chest side will receive only standard of care and normal wound dressing.
  Interventions: Device: Brijjit® BP100-6 and BP-75; Other: Control: Standard of care and normal wound dressing

INTERVENTIONS:
Device: Brijjit® BP100-6 and BP-75 — Brijjit® BP-100 and BP-75 are a non-invasive, flexible devices that acts as a force modulating tissue bridge (FMTB) to aid in wound healing. BP-100 and BP-75 simply refer to different sizes of the Brijjit device.
Other: Control: Standard of care and normal wound dressing — The control chest side will receive only standard of care and normal wound dressing.

SUMMARY:
The goal of this randomized, prospective, interventional clinical trial is to evaluate the use of Brijjit® in reducing the incidence of hypertrophic scarring in individuals undergoing gender-affirming bilateral double incision mastectomies at a single-institution, single-surgeon site (Esther A. Kim, MD). Patients will serve as a self-control (one side of the chest receives intervention, the other serves as a control). Primary endpoints include scar appearance and quality. Secondary endpoints include patient perception of the scar using the Patient and Observer Scar Assessment Scale (POSAS).

Participants will be taught how to apply Brijjit® at home if any units fall off before 6 weeks postop.

DETAILED DESCRIPTION:
The hypothesis of this study is that the use of Brijjit® Force-Modulating Tissue Bridge devices will reduce the incidence of hypertrophic scarring as measured by objective and subjective factors compared to no intervention following gender-affirming double incision mastectomy. Patients will serve as self-controls (one side of the chest will receive the intervention, the other will not). Consistent use of silicone-based tape, the current gold standard for wound care, will be encouraged on the control side of the chest.

We hypothesize that applying FMTBs to surgical incisions will improve scar outcomes by limiting pro-fibrotic signaling and promoting optimal wound healing. Should our hypotheses be proven, this study will provide a compelling reason to implement Brijjit therapy into standard clinical practice as a non-invasive preventative measure to improve scar outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19
2. Undergoing double incision gender affirming mastectomy
3. Ability to adhere to Brijjit therapy after surgery
4. Willing to return for follow-up visits and undergo study evaluations

Exclusion Criteria:

1. History of keloid formation
2. Radiation therapy history
3. Prior surgeries of the chest or breast
4. History or use following prescription medications: 1) accutane within the past year. 2) chronic systemic steroids
5. Active smoker
6. Disorder known to negatively affect wound healing (autoimmune, connective tissue, uncontrolled diabetes)
7. Any other condition determined by PI to preclude subject from joining study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identifying as transgender, gender expansive, or non-binary
Enrollment: 78 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Presence of Hypertrophic Scarring | 6 weeks postop
  Presence or Absence of HTS: HTS defined as a raised, firm fibrotic lesion that develops within the boundaries of surgical incision with a height cutoff of >/= 1mm. Binary yes or no outcome.
Presence of Hypertrophic Scarring | 3 months postop
  Presence or Absence of HTS: HTS defined as a raised, firm fibrotic lesion that develops within the boundaries of surgical incision with a height cutoff of >/= 1mm. Binary yes or no outcome.
Presence of Hypertrophic Scarring | 6 months postop
  Presence or Absence of HTS: HTS defined as a raised, firm fibrotic lesion that develops within the boundaries of surgical incision with a height cutoff of >/= 1mm. Binary yes or no outcome.
Presence of Hypertrophic Scarring | 1 year postop
  Presence or Absence of HTS: HTS defined as a raised, firm fibrotic lesion that develops within the boundaries of surgical incision with a height cutoff of >/= 1mm. Binary yes or no outcome.
Scar Characteristics | 6 weeks postop
  Qualitative description of scar: Scar color, pigmentation, texture, description (flat, thin, depressed, spread, raised)
Scar characteristics | 3 months postop
  Qualitative description of scar: Scar color, pigmentation, texture, description (flat, thin, depressed, spread, raised)
Scar Characteristics | 6 months postop
  Qualitative description of scar: Scar color, pigmentation, texture, description (flat, thin, depressed, spread, raised)
Scar Characteristics | 1 year postop
  Qualitative description of scar: Scar color, pigmentation, texture, description (flat, thin, depressed, spread, raised)
Scar Dimensions | 6 weeks postop
  Scar Scar length, width and thickness measured in cm. If HTS present: Length of HTS and incision ratio Location of HTS: Medial, Middle, or Lateral. Measured distance from sternum.
Scar Dimensions | 3 months postop
  Scar Scar length, width and thickness measured in cm. If HTS present: Length of HTS and incision ratio Location of HTS: Medial, Middle, or Lateral. Measured distance from sternum.
Scar Dimensions | 6 months postop
  Scar Scar length, width and thickness measured in cm. If HTS present: Length of HTS and incision ratio Location of HTS: Medial, Middle, or Lateral. Measured distance from sternum.
Scar Dimensions | 1 year postop
  Scar Scar length, width and thickness measured in cm. If HTS present: Length of HTS and incision ratio Location of HTS: Medial, Middle, or Lateral. Measured distance from sternum.

SECONDARY OUTCOMES:
Patient Perception of Scar | 6 weeks postop
  Use the Patient and Observer Scar Assessment Scale (POSAS): A validated, widely used questionnaire consisting of both patient and observer scales regarding scar appearance, physical symptoms (e.g. pain, pruritus), and overall patient satisfaction. This scale allows for scores ranging from 1-10, with higher scores meaning a worse outcome. Patients will be given this survey in clinic, but will be given the option of completing it electronically at home.
Patient Perception of Scar | 3 months postop
  Use the Patient and Observer Scar Assessment Scale (POSAS): A validated, widely used questionnaire consisting of both patient and observer scales regarding scar appearance, physical symptoms (e.g. pain, pruritus), and overall patient satisfaction. This scale allows for scores ranging from 1-10, with higher scores meaning a worse outcome. Patients will be given this survey in clinic, but will be given the option of completing it electronically at home.
Patient Perception of Scar | 6 months postop
  Use the Patient and Observer Scar Assessment Scale (POSAS): A validated, widely used questionnaire consisting of both patient and observer scales regarding scar appearance, physical symptoms (e.g. pain, pruritus), and overall patient satisfaction. This scale allows for scores ranging from 1-10, with higher scores meaning a worse outcome. Patients will be given this survey in clinic, but will be given the option of completing it electronically at home.
Patient Perception of Scar | 1 year postop
  Use the Patient and Observer Scar Assessment Scale (POSAS): A validated, widely used questionnaire consisting of both patient and observer scales regarding scar appearance, physical symptoms (e.g. pain, pruritus), and overall patient satisfaction. This scale allows for scores ranging from 1-10, with higher scores meaning a worse outcome. Patients will be given this survey in clinic, but will be given the option of completing it electronically at home.

CONTACTS AND LOCATIONS:
Overall Officials: Esther A Kim, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- UCSF Department of Plastic & Reconstructive Surgery, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panton J, Vingan N, Barillas J, Akgul Y, Lazzarini A, Coroneos CJ, Amirlak B, Kenkel J, Culver A. Postoperative Mechanomodulation Decreases T-Junction Dehiscence After Reduction Mammaplasty: Early Scar Analysis From a Randomized Controlled Trial. Aesthet Surg J. 2023 Nov 16;43(12):NP1033-NP1048. doi: 10.1093/asj/sjad269. PMID 37606245
- [Background] Cao G, Ye M, Wang H, Liu Y, Li M. The Role of Biomechanical Forces in the Formation and Treatment of Pathological Scars. Clin Cosmet Investig Dermatol. 2024 Nov 13;17:2565-2571. doi: 10.2147/CCID.S496253. eCollection 2024. PMID 39559183
- See also: Tension Reduction With Force Modulating Tissue Bridges Reduces Wound Formation in Elective Breast Surgery — https://pubmed.ncbi.nlm.nih.gov/37652052/
- See also: Mechanomodulation of Wound Healing: Current Perspectives and Future Directions — https://doi.org/10.1016/j.jid.2021.10.003
- See also: Silicone in Scar Prevention and Treatment: A Review of Current Evidence — https://doi.org/10.1016/j.bjps.2015.09.013
- See also: Mechanical Forces in Cutaneous Wound Healing: Emerging Therapies to Minimize Scar Formation — https://pmc.ncbi.nlm.nih.gov/articles/PMC5792236/